CLINICAL TRIAL: NCT00235157
Title: Palmaz Genesis Peripheral Stainless Steel Balloon Expandable Stent, Comparing a Sirolimus Coated Versus an Uncoated Stent in REnal Artery Treatment.
Brief Title: A Comparison of Coated and Uncoated Stents in Renal Artery Treatment.
Acronym: GREAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Director Clinical Affairs, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EE01-01
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Sirolimus-eluting Palmaz Genesis peripheral stent
  Interventions: Device: Sirolimus-eluting Palmaz Genesis peripheral stent

INTERVENTIONS:
Device: Sirolimus-eluting Palmaz Genesis peripheral stent — treatment of renal artery stenosis with a renal stent
  Other Names: Palmaz Genesis Stent

SUMMARY:
The primary objective of this study is to compare the safety and performance of the Palmaz Genesis™ balloon expandable stent, with or without sirolimus coating in the treatment of renal artery stenosis, measured at 6 months follow up via angiography.

DETAILED DESCRIPTION:
Multi-center, prospective, controlled, non-randomized investigational feasibility study. One hundred (100) patients with de novo or restenotic renal artery lesions consisting of >= 50% stenosis and reference vessel of >= 4.0 to <= 8.0 mm in diameter will be sequentially included, 50 without sirolimus coating, followed by 50 with sirolimus coating Palmaz GenesisTM. Patients will be followed for 24 months post-procedure, with all patients having clinical assessments at discharge, 1,6, 12 and 24 months. This study will be conducted at twelve investigational sites.

It is anticipated that the total length of time required to complete the study will be 46 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for renal artery revascularization of atherosclerotic renal artery stenosis >=50% as measured by operator or estimated original vessel diameter, based on healthy vessel segment and contralateral side.
2. The reference vessel renal artery must be >= 4mm and <= 8 mm by visual estimate.
3. The patient must have a baseline serum creatinine of <= 5.0 mg/dl.

Exclusion Criteria:

1. Total occlusion of the renal artery.
2. Lesions which would require more than 2 stents.
3. Lesions which are in arteries to transplanted or bypassed kidneys.
4. Abdominal aortic aneurysm > 4.0 cm in diameter.
5. Patients with ASA classification >=4.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-11; Primary Completion 2002-11 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
assessment of the angiographical in-stent minimal lumen diameter | 6-months follow up

SECONDARY OUTCOMES:
clinical primary patency | discharge, 1, 6 and 12 months post-procedure
procedural success | post-procedure
worsening renal function | 30 days, 6 months, 12 months
change in blood pressure measurement | 30 days, 6 months, 12 months
significant embolic events causing end-organ damage | 30 days, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zähringer, MD, Principal Investigator — Universitätskliniken Köln; Marc Sapoval, MD, Principal Investigator — Hopital Européen Georges Pompidou; Peter M Pattynama, MD, Principal Investigator — Erasmus MC Rotterdam
Locations (3):
- Hopital Européen Georges Pompidou, Paris, France
- Universitätskliniken Köln, Cologne, Germany
- Erasmus MC Rotterdam, Rotterdam, Netherlands

REFERENCES:
- [Result] Zahringer M, Sapoval M, Pattynama PM, Rabbia C, Vignali C, Maleux G, Boyer L, Szczerbo-Trojanowska M, Jaschke W, Hafsahl G, Downes M, Beregi JP, Veeger NJ, Stoll HP, Talen A. Sirolimus-eluting versus bare-metal low-profile stent for renal artery treatment (GREAT Trial): angiographic follow-up after 6 months and clinical outcome up to 2 years. J Endovasc Ther. 2007 Aug;14(4):460-8. doi: 10.1177/152660280701400405. PMID 17696619